CLINICAL TRIAL: NCT05642819
Title: Routine Evaluation of People Living With Cancer - Surgery
Brief Title: REVOLUTION Surgery (REVOLUTION Surgery)
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC22098
Record Dates: First submitted 2022-09-15; First posted 2022-12-08 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Cachexia; Oesophageal Cancer; Gastric Cancer; Pancreatic Cancer; Colorectal Cancer
MeSH Terms: conditions — Cachexia; Esophageal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood samples - approximately 40mls. Urine samples - approximately 20mls. Muscle samples - small sample Fat samples - small sample Tumour samples - small sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer Resection: * Patients with cancer (clinical, histological, cytological or radiological evidence) planned for surgical resection of a malignancy of the oesophagus, stomach, pancreas, colon, or rectum
  * Aged 18-years and over
  * Able to give written informed consent
- Healthy Controls: * Patients identified at surgical clinic as being planned for an open abdominal operation for a non-inflammatory, benign condition (e.g. donor nephrectomy)
  * Aged 18-years and over
  * Able to give written informed consent

SUMMARY:
Some people with cancer suffer from muscle wasting, lose weight and feel tired. This process, termed cachexia, is a significant problem and can lead to a reduction in both quality and quantity of life.

Cachexia is caused by interactions between the tumour and the patient. Historically, it was considered to be a purely end-stage phenomenon of advanced cancer, however, it is now known that early signs of cachexia can even influence the outcomes of patients with potentially curative pathology, including those planned for a surgical resection.

This study aims to collect information, from patients who are at risk of cachexia, about body composition, physical activity, quality of life and the body's immune response to cancer. Previously these measures have been most frequently studied in isolation, or at one single time-point, and are therefore likely to give an incomplete picture. A more holistic characterisation of surgical patients at risk of cancer cachexia, across their treatments, is currently lacking.

Participants with cancer will be recruited to the study from surgical services in the United Kingdom (UK). A small number of 'control' patients without cancer, who are undergoing surgery for a benign condition, will also be recruited for comparison. Those recruited will have their height and weight measured, answer questionnaires about quality of life, undergo assessment of their physical function and levels of activity, have blood taken to analyse markers of inflammation and have their body composition measured by a variety of methods. A subgroup of patients will also undergo an additional magnetic resonance imaging (MRI) scan of their abdomen and thighs. At the time of their operation, participants will also have small biopsies of muscle, fat, tumour and urine taken for biochemical analysis. Patients with cancer, will be asked to return for three follow up appointments during the year after their operation where these assessments will be repeated.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria (Cancer Resection)

* Patients with cancer (Clinical, histological, cytological or radiological evidence) planned for surgical resection of a malignancy of the oesophagus, stomach, pancreas, colon, or rectum
* Aged 18-years and over
* Able to give written informed consent

Inclusion Criteria (Healthy Controls)

* Patients identified at surgical clinic as being planned for an open abdominal operation for a non-inflammatory, benign condition (e.g. donor nephrectomy)
* Aged 18-years and over
* Able to give written informed consent

Exclusion Criteria:

* Any concomitant medical or psychiatric problems which, in the opinion of the investigator, would increase the risk of complication for the participant and/or investigator
* Presence of a concomitant inflammatory (e.g., rheumatoid arthritis, inflammatory bowel disease) or muscle wasting condition other than cancer
* Participants who are pregnant, suffer from claustrophobia or with implanted medical devices (e.g., cardiac pacemaker, metallic foreign bodies, aneurysm clip) would not be able to undergo the additional multiparametric magnetic resonance imaging (MRI)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients planned for surgical resection of a gastrointestinal tract cancer, at risk of cancer cachexia, recruited from surgical services in the UK.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Longitudinal changes in weight | Measured at baseline, following completion of any neo-adjuvant anti-cancer therapy, 6 (+/- 2) weeks, 6 (+/- 1) months and 12 (+/- 1) months following surgical resection
  Longitudinal changes in weight (kg) - combined with height (m) to report body mass index (BMI) (kg/m2)
Longitudinal changes in computed tomography (CT) body composition (muscle quantity) | Measured at staging CT scan, at repeat scan following any neoadjuvant anti-cancer therapies and at follow-up scans following surgical resection / adjuvant anti-cancer therapies and other scans up to 1 year post surgical resection
  Longitudinal changes in cross-sectional area (cm2) and volume (cm3) of skeletal muscle and radiodensity of skeletal muscle, subcutaneous fat, visceral fat and intra-muscular adipose tissue.
Longitudinal changes in CT body composition (muscle radiodensity) | Measured at staging CT scan, at repeat scan following any neoadjuvant anti-cancer therapies and at follow-up scans following surgical resection / adjuvant anti-cancer therapies and other scans up to 1 year post surgical resection
  Longitudinal changes in radiodensity (HU - Hounsfield units) of skeletal muscle
Longitudinal changes in CT body composition (fat quantity) | Measured at staging CT scan, at repeat scan following any neoadjuvant anti-cancer therapies and at follow-up scans following surgical resection / adjuvant anti-cancer therapies and other scans up to 1 year post surgical resection
  Longitudinal changes in cross-sectional area (cm2) and volume (cm3) of subcutaneous and visceral adipose tissue
Longitudinal changes in CT body composition (fat radiodensity) | Measured at staging CT scan, at repeat scan following any neoadjuvant anti-cancer therapies and at follow-up scans following surgical resection / adjuvant anti-cancer therapies and other scans up to 1 year post surgical resection
  Longitudinal changes in radiodensity (HU - Hounsfield units) of subcutaneous and visceral adipose tissue
Longitudinal changes in systemic inflammation | Measured at baseline, following completion of any neo-adjuvant anti-cancer therapy, 6 (+/- 2) weeks, 6 (+/- 1) months and 12 (+/- 1) months following surgical resection
  Longitudinal changes in serum levels of pro-inflammatory cytokines and other markers of systemic inflammation
Longitudinal changes in physical activity | Measured at baseline, following completion of any neo-adjuvant anti-cancer therapy, 6 (+/- 2) weeks, 6 (+/- 1) months and 12 (+/- 1) months following surgical resection
  A personal activity monitor (FitBit) will be worn for the next eight days to assess step count and time of physical activity
Longitudinal changes in muscle function | Measured at baseline, following completion of any neo-adjuvant anti-cancer therapy, 6 (+/- 2) weeks, 6 (+/- 1) months and 12 (+/- 1) months following surgical resection
  The 'timed up and go' test will be assessed for all participants as an estimate of lower limb muscle function
Longitudinal changes in muscle strength | Measured at baseline, following completion of any neo-adjuvant anti-cancer therapy, 6 (+/- 2) weeks, 6 (+/- 1) months and 12 (+/- 1) months following surgical resection
  Isometric knee extension will be assessed for patients undergoing a multiparametric MRI as an estimate of quadriceps strength. This will be done using a hand-held dynamometer.
Longitudinal changes in risk of nutritional deficit | Measured at baseline, following completion of any neo-adjuvant anti-cancer therapy, 6 (+/- 2) weeks, 6 (+/- 1) months and 12 (+/- 1) months following surgical resection
  Patient Generated Subjective Global Assessment Short Form ('PG-SGA-SF') questionnaires will be used to assess symptom burden and quality of life measures, specifically regarding nutritional risk in catabolic conditions
Longitudinal changes in quality of life (physical, psychological and social function in patients with cancer) | Measured at baseline, following completion of any neo-adjuvant anti-cancer therapy, 6 (+/- 2) weeks, 6 (+/- 1) months and 12 (+/- 1) months following surgical resection
  European Organisation For Research And Treatment Of Cancer Quality of Life Questionnaire C30 ('EORTC-QLQ-C30') questionnaires will be used to assess symptom burden and general quality of life
Longitudinal changes in symptom burden, function and general quality of life in patients with anorexia / cachexia) | Measured at baseline, following completion of any neo-adjuvant anti-cancer therapy, 6 (+/- 2) weeks, 6 (+/- 1) months and 12 (+/- 1) months following surgical resection
  Functional Assessment of Anorexia / Cachexia Therapy ('FAACT') questionnaires will be used to assess symptom burden, quality of life and function
Longitudinal tissue-level changes in fat content | Muscle biopsies will be taken at the time of surgical resection. Where participants are amenable, additional repeat needle biopsies of the quadriceps muscle will be performed at follow-up appointments 6 (+/- 1) months and 12 (+/- 1) months post surgery
  Longitudinal changes in tissue level changes associated with cachexia, such as fat content of skeletal muscle
Longitudinal tissue-level changes in collagen content | Muscle biopsies will be taken at the time of surgical resection. Where participants are amenable, additional repeat needle biopsies of the quadriceps muscle will be performed at follow-up appointments 6 (+/- 1) months and 12 (+/- 1) months post surgery
  Longitudinal changes in tissue level changes associated with cachexia, such as collagen content of skeletal muscle
Longitudinal tissue-level changes in protein content | Muscle biopsies will be taken at the time of surgical resection. Where participants are amenable, additional repeat needle biopsies of the quadriceps muscle will be performed at follow-up appointments 6 (+/- 1) months and 12 (+/- 1) months post surgery
  Longitudinal changes in tissue level changes associated with cachexia, such as protein content of skeletal muscle
Evaluation of multiparametric magnetic resonance imaging (MRI) in cachexia | MRI scan performed pre-operatively
  Evaluation of multiparametric MRI as a novel method for estimation of skeletal muscle mass and fat-infiltration across cachectic and weight-stable patients with cancer

SECONDARY OUTCOMES:
Correlation of multiparametric magnetic resonance imaging (MRI) and tissue-level changes | MRI scan performed pre-operatively, tissue samples collected at the point of surgical resection.
  Correlation of multiparametric MRI estimates of skeletal muscle mass and fat infiltration with CT image derived analyses and tissue level changes in fat, collagen and protein content of skeletal muscle.
Correlation of multiparametric magnetic resonance imaging (MRI) and changes in physical function | MRI scan and assessments of physical function & muscle strength performed pre-operatively.
  Evaluation of the relationship between physical function & muscle strength (as assessed by personal activity monitor (FitBit), 'timed up and go' test and isometric knee extension using a hand-held dynamometer) and multiparametric MRI assessment of thigh muscle quantity.

CONTACTS AND LOCATIONS:
Overall Officials: Richard JE Skipworth, MD FRCS, Principal Investigator — University of Edinburgh / NHS Lothian
Locations (1):
- University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
To be confirmed